CLINICAL TRIAL: NCT03859375
Title: Number of Necessary Paints of Preoperative Skin Disinfection to Prevent Surgical Site Infections; PAINTS Study
Brief Title: Number of Necessary Paints of Preoperative Skin Disinfection to Prevent Surgical Site Infections
Acronym: PAINTS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02292; me18Widmer2
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Surgical Site Infection
Keywords: Colony forming units; preoperative skin disinfection; microbial skin counts
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2 paints of skin disinfectants: Standard microbial swabs (eSWAB) to do microbial skin counts in the disinfection area after paints of skin disinfectants will be taken by the operating room-nurses prior to skin disinfection and after paint two of a predefined area of the skin.
  Interventions: Other: microbial skin counts in the disinfection area after paints of skin disinfectants
- 3 paints of skin disinfectants: Standard microbial swabs (eSWAB) to do microbial skin counts in the disinfection area after paints of skin disinfectants will be taken by the operating room-nurses prior to skin disinfection and after paint three of a predefined area of the skin.
  Interventions: Other: microbial skin counts in the disinfection area after paints of skin disinfectants

INTERVENTIONS:
Other: microbial skin counts in the disinfection area after paints of skin disinfectants — microbial skin counts in the disinfection area after 2 and 3 paints of skin disinfectants (chlorhexidine in alcohol [CHX] and povidone iodine in alcohol [PI])

SUMMARY:
This observational study investigates whether 3 paints are superior compared to 2 paints in reducing microbial skin counts in the disinfection area of cardiac and abdominal surgery patients.

DETAILED DESCRIPTION:
Surgical site infection (SSI) remain the most common nosocomial infection in surgical departments. Preparation of the skin with disinfectants belongs to the standard of care prior to any surgical intervention but disinfection practices are heterogeneous across different hospitals and countries. Although the efficacy and effectiveness of preoperative surgical site preparation is dependent on both the antiseptic agent used and the application method, it is unclear how many paints of an antiseptic are needed to ensure adequate infection protection.

An adequately powered study including different standard antiseptic agents (i.e. chlorhexidine in alcohol (CHX) and povidone iodine in alcohol (PI)) is therefore required to compare the protective effect of different numbers of paints.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective cardiac surgery at the study site
* Adult patients undergoing elective abdominal surgery at the study site
* Provision of informed consent

Exclusion Criteria:

* Pregnancy reported by patient
* Emergency (non-elective) surgical interventions
* Contraindications to the use of either one of the compounds: Alcoholic CHX; Alcoholic PI
* Skin or other hypersensitivity reactions during the disinfection process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac or abdominal (colorectal surgery, cholecystectomy) interventions at the University Hospital of Basel will be eligible for this study unless meeting exclusion criteria
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Change in microbial skin counts (number of Colony forming Units (CFU)) | prior to skin disinfection (T0) and after paint two (T1, approx. after 2 minutes) and after paint three (T2; approx. after 3 minutes) before start of surgery
  Change in microbial skin counts (CFU) after 3 paints as compared to 2 paints

SECONDARY OUTCOMES:
Proportion of patients with microbial skin counts of 0 CFU after 3 paints as compared to 2 paints | after paint two (T1, approx. after 2 minutes) and after paint three (T2; approx. after 3 minutes) before start of surgery
  Proportion of patients with microbial skin counts of 0 CFU after 3 paints as compared to 2 paints
Proportion of patients with insufficient reduction of microbial skin counts (i.e. log reduction of CFU <2) after 2 paints | after paint two (T1, approx. after 2 minutes)
  Proportion of patients with insufficient reduction of microbial skin counts (i.e. log reduction of CFU <2) after 2 paints

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Widmer, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland